CLINICAL TRIAL: NCT03397082
Title: Topic Use of Lidocaine Gel Plus Paracervical Blockade vs. Paracervical Blockade Alone for Pain Control During Endouterine Manual Aspiration: A Randomized Controlled Trial
Brief Title: Topic Cervical Anesthesia for Pain Control During Endouterine Manual Aspiration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saint Thomas Hospital, Panama (Other)
Responsible Party: Principal Investigator, Osvaldo A. Reyes T., Coordinator Research Department, Saint Thomas Hospital, Panama
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mhst2014-13
Record Dates: First submitted 2018-01-02; First posted 2018-01-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Pain
Keywords: Endouterine manual aspiration; Paracervical blockade; Lidocaine gel
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine + Paracervical blockade (Experimental): 5 minutes previous to endouterine manual aspiration, 5mL of lidocaine gel was applied plus standard paracervical blockade.
  Interventions: Drug: Lidocaine gel
- Placebo + paracervical blockade (Placebo Comparator): 5 minutes previous to endouterine manual aspiration, standard paracervical blockade was applied plus placebo gel (KY).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lidocaine gel — 5mL of lidocaine gel applied topically to cervix previous to clamping and paracervical blockade.
  Arms: Lidocaine + Paracervical blockade
Drug: Placebo — 5mL of sterile gel applied topically to cervix previous to clamping and paracervical blockade.
  Arms: Placebo + paracervical blockade

SUMMARY:
To compare the effectiveness of lidocaine gel plus paracervical blockade vs. Paracervical blockade alone in the management of pain during endouterine manual aspiration.

ELIGIBILITY:
Inclusion Criteria:

* Need for a endouterine manual aspiration (incomplete abortion or gynecological bleeding).

Exclusion Criteria:

* Allergy to lidocaine.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2014-09-30 (Actual); Study Completion 2014-12-01 (Actual)

PRIMARY OUTCOMES:
Global evaluation of pain | 5 minutes post procedure
  Visual scale of pain evaluation

SECONDARY OUTCOMES:
Adverse reaction | 5 minutes post procedure
  Presence of adverse effects to the drug used (lidocaine gel)

CONTACTS AND LOCATIONS:
Overall Officials: Osvaldo Reyes, Md, Study Director — Saint Thomas Maternity Hospital; Ariel Veces, Principal Investigator — Saint Thomas Maternity Hospital
Locations (1):
- Saint Thomas Maternity Hospital, Panama City, Panama

IPD SHARING:
Plan to Share IPD: No